CLINICAL TRIAL: NCT01807494
Title: Direct Anterior Versus Posterior Total Hip Arthroplasty Surgical Approaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New Lexington Clinic (Other)
Collaborators: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCO.2012.05
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posterior approach (Active Comparator): Subjects in this group will total hip replacement performed with a posterior surgical approach and total hip replacement components.
  Interventions: Device: Total hip replacement components
- Anterior Approach (Active Comparator): Subjects in this group will have total hip replacement performed with a direct anterior surgical approach and total hip replacement components.
  Interventions: Device: Total hip replacement components

INTERVENTIONS:
Device: Total hip replacement components — All patients will receive the same implants
  Other Names: Femoral component will be the Biomet Taperloc Complete and the acetabular component will be the Biomet Ringloc+

SUMMARY:
Hip replacement is a common surgical procedure performed to relieve the pain and disability. In general, the surgery consists of replacing the diseased or damaged joint surfaces of the hip with metal and plastic components shaped to allow continued motion of the hip. Surgeons may perform this operation in several different ways. The purpose of this study is to compare two different methods of performing total hip replacement. The investigators hypothesize that subjects treated with the anterior approached may show improved function during the early postoperative period, but that no differences in pain or function will be present after the first postoperative year.

In this study, patients that have elected to have hip replacement and consented to participate in the study will be randomized to have his or her hip replaced using one of two surgical techniques. Subjects will be randomized to be implanted using either an anterior or posterior approach. With the anterior approach, the study surgeon will use an incision that is on the front of the hip, and with the posterior approach, the incision will be more on the backside of your hip. The study surgeon has done more than 300 total hip replacements with both of these techniques.

A baseline assessment will be conducted before hip replacement surgery that includes x-rays, functional tasks like getting up from a chair and stepping down a step, and three questionnaires about the hip, the subject's general health, and how well the subject is able to function. Also, subjects will be required to return to the clinic at several time points after surgery for follow-up visits. Follow-up visits will include hip assessments and questionnaires, as well as follow-up hip x-rays. The follow-up visits will be 6 weeks, 3 months, 1 year, 2 years, 5 years, 7 years, and 10 years after hip replacement surgery. These follow-up visits are part of the study surgeon's normal routine for hip replacement patients, and are not extra visits as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 85
* End stage hip joint degeneration
* Has elected to undergo primary total hip arthroplasty

Exclusion Criteria:

* Undergoing revision arthroplasty
* Inflammatory or rheumatoid arthritis
* Patients with confounding medical conditions that are not expected to survive for the duration of follow-up (10 years)
* Body Mass Index greater than 40 kg/m2
* Age < 18 or > than 85
* Previous ipsilateral hip surgery including arthroscopic procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Time to discontinued use of an assistive ambulatory device (cane or walker) | 6 week postoperative follow-up

SECONDARY OUTCOMES:
modified Harris Hip Score | Preoperative (no more than 3 months before surgery), and at 6-week, 12-week, 1-, 2-, 5-, 7-, and 10-year follow-ups
SF-12 | Preoperative (no more than 3 months before surgery), and at 6-week, 12-week, 1-, 2-, 5-, 7-, and 10-year follow-ups
Lower Extremity Functional Score | Preoperative (no more than 3 months before surgery), and at 6-week, 12-week, 1-, 2-, 5-, 7-, and 10-year follow-ups
Functional force testing | Preoperative (no more than 3 months before surgery), and at 6-week, 12-week, 1-, 2-, 5-, 7-, and 10-year follow-ups
  Testing to objectively quantify subject function when rising from a chair and descending stairs
implant survivorship | 1-, 2-, 5-, 7-, and 10-year follow-ups
Length of hospital stay | Collected during the hospital stay (usually 1 to 5 days)
Operative time | Intra-operative
Number of patients that require blood transfusion | Intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Christensen, MD, Principal Investigator — Lexington Clinic
Locations (1):
- Lexington Clinic, Lexington, Kentucky, United States